CLINICAL TRIAL: NCT06686563
Title: Audiovisual Stimulation in Elderly (Older Adults?): Effects on Cognition, Depressive Symptoms, and Dual Motor-Cognitive Tasks - a RCT
Brief Title: WAVE: AudioVisual Stimulation Enhances Cognitive, Mental and Physical Health in Elderly
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Maria Paço (Other)
Collaborators: Universidade do Sul de Santa Catarina (Other Government)
Responsible Party: Sponsor-Investigator, Maria Paço, PhD, Cooperativa de Ensino Superior, Politécnico e Universitário
Organization: Cooperativa de Ensino Superior, Politécnico e Universitário (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WAVE_56/CE-IPSN/2023
Record Dates: First submitted 2024-07-17; First posted 2024-11-13 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Mild Cognitive Impairment
Keywords: Cognitive decline; Depressive symptoms; Audiovisual stimulation; Inflammaging; Older adults
MeSH Terms: conditions — Cognitive Dysfunction; Depression

STUDY DESIGN:
Intervention Model Description: A double-blind randomized controlled clinical trial will be conducted with 48 elderly volunteers from a daycare center in Famalicão. After an initial cognitive screening (MoCA), assessment of depressive symptoms (GDS-15), agility and functional balance (TUG), and chronic inflammatory conditions (blood analysis), participants will be randomly assigned to a group (IG: intervention group; CG: control group). Participants in the CG will be stimulated with theta frequency (4-7 Hz), while participants in the IG will be stimulated with gamma frequency (39-42 Hz). For both groups, the frequency of the intervention will be 5 times a week, with the AVNS being used twice a week for 20 minutes (a minimum of 20 sessions - 8 to 12 weeks) and the other 3 days being spent at home with 20 minutes of audio frequency stimulation at the appropriate frequency (GC: theta, GI: gamma). After this period, all participants will be re-evaluated.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants in the IG will be stimulated with gamma frequency (39-42 Hz). The frequency of the intervention will be 5 times a week, with the AVNS being used twice a week for 20 minutes (a minimum of 20 sessions - 8 to 12 weeks) and the other 3 days being spent at home with 20 minutes of audio frequency stimulation.
  The participants will be assessed (regarding the outcomes previously described) at the baseline and reassessed after 3 months.
  Interventions: Other: Intervention Group: Gamma stimulation
- Control Group (Active Comparator): Participants in the CG will be stimulated with theta frequency (4-7 Hz). The frequency of the intervention will be 5 times a week, with the AVNS being used twice a week for 20 minutes (a minimum of 20 sessions - 8 to 12 weeks) and the other 3 days being spent at home with 20 minutes of audio frequency stimulation.
  The participants will be assessed (regarding the outcomes previously described) at the baseline and reassessed after 3 months.
  Interventions: Other: Control Group: Theta stimulation

INTERVENTIONS:
Other: Intervention Group: Gamma stimulation — Participants in this group be stimulated with gamma frequency (39-42 Hz). The frequency of the intervention will be 5 times a week, with the AVNS being used twice a week for 20 minutes (a minimum of 20 sessions - 8 to 12 weeks) and the other 3 days being spent at home with 20 minutes of audio frequency stimulation.
  Arms: Intervention Group
Other: Control Group: Theta stimulation — Participants in this group will be stimulated with theta frequency (4-7 Hz). The frequency of the intervention will be 5 times a week, with the AVNS being used twice a week for 20 minutes (a minimum of 20 sessions - 8 to 12 weeks) and the other 3 days being spent at home with 20 minutes of audio frequency stimulation.
  Arms: Control Group

SUMMARY:
The goal of this randomized controlled trial is to 1) carry out a screening of cognitive function, depressive symptoms, agility and functional balance and chronic inflammatory conditions in older adults; 2) analyze the influence of AVNS on cognitive function, depressive symptoms, agility and functional balance and chronic inflammatory conditions in older adults.

The main question it aims to answer is: "Does AVNS have influence on cognitive function, depressive symptoms, agility and functional balance and chronic inflammatory conditions in older adults ". Participants will be randomly assigned to a control group or to a intervention group, where they will use AVNS to see if influences the above mentioned outcomes, compared to the no intervention (control) group.

DETAILED DESCRIPTION:
Mild Cognitive Impairment (MCI) can be defined as a pre-dementia symptom and, when associated with aging, characterizes individuals with cognitive decline below the level of dementia. This decline, which can begin as early as 45 years of age, leads to impairments in memory, learning, language, orientation, and executive functions, which are more visible from the sixth decade of life onwards, with a risk of reduced autonomy and independence, and is seen by researchers as the first stage of a process of loss. This loss is progressive, lasting several years and resulting in MCI, characterized by objective cognitive loss, which does not yet compromise autonomy but has a conversion rate to dementia of 10% per year. Cognitive decline can be accompanied by increased depressive symptoms and decreased functional capacity and is related to inflammatory conditions, described in the literature as "inflammaging". Studies with beat stimulation have shown benefits in different important outcomes of cognitive function and depression. Thus, audiovisual neurostimulation (AVNS) is a possible non-pharmacological treatment that might have a direct influence on the brain wave patterns, altered in MCI and depression, modulating these specific wave frequencies to functional patterns similar to those found in healthy individuals. Having this, it can also influence agility and functional balance and reduce chronic inflammatory conditions.

ELIGIBILITY:
Inclusion Criteria:

* Know how to read and write

Exclusion Criteria:

-

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Cognitive screening | From enrollment to the end of intervention
  Montreal Cognitive Assessment (MoCA)
Performance of the dual motor-cognitive task | From enrollment to the end of intervention
  Timed Up and Go (TUG)
Blood biomarkers for chronic inflammatory conditions | From enrollment to the end of intervention

SECONDARY OUTCOMES:
Depressive symptoms | From enrollment to the end of intervention
  Geriatric Depressive Scale 15 items (GDS-15)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Quialheiro, PhD, Principal Investigator — Cooperativa de Ensino Superior, Politécnico e Universitário
Locations (1):
- Cooperativa Ensino Superior Politécnico e Universitário, Gandra, Paredes, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Albert MS, DeKosky ST, Dickson D, Dubois B, Feldman HH, Fox NC, Gamst A, Holtzman DM, Jagust WJ, Petersen RC, Snyder PJ, Carrillo MC, Thies B, Phelps CH. The diagnosis of mild cognitive impairment due to Alzheimer's disease: recommendations from the National Institute on Aging-Alzheimer's Association workgroups on diagnostic guidelines for Alzheimer's disease. Alzheimers Dement. 2011 May;7(3):270-9. doi: 10.1016/j.jalz.2011.03.008. Epub 2011 Apr 21. PMID 21514249
- [Background] Singh-Manoux A, Kivimaki M, Glymour MM, Elbaz A, Berr C, Ebmeier KP, Ferrie JE, Dugravot A. Timing of onset of cognitive decline: results from Whitehall II prospective cohort study. BMJ. 2012 Jan 5;344:d7622. doi: 10.1136/bmj.d7622. PMID 22223828
- [Background] Ramos LR, Simoes EJ, Albert MS. Dependence in activities of daily living and cognitive impairment strongly predicted mortality in older urban residents in Brazil: a 2-year follow-up. J Am Geriatr Soc. 2001 Sep;49(9):1168-75. doi: 10.1046/j.1532-5415.2001.49233.x. PMID 11559375
- [Background] Yesavage JA, O'Hara R, Kraemer H, Noda A, Taylor JL, Ferris S, Gely-Nargeot MC, Rosen A, Friedman L, Sheikh J, Derouesne C. Modeling the prevalence and incidence of Alzheimer's disease and mild cognitive impairment. J Psychiatr Res. 2002 Sep-Oct;36(5):281-6. doi: 10.1016/s0022-3956(02)00020-1. PMID 12127595
- [Background] Morris JC, Storandt M, Miller JP, McKeel DW, Price JL, Rubin EH, Berg L. Mild cognitive impairment represents early-stage Alzheimer disease. Arch Neurol. 2001 Mar;58(3):397-405. doi: 10.1001/archneur.58.3.397. PMID 11255443
- [Background] Franceschi C, Garagnani P, Parini P, Giuliani C, Santoro A. Inflammaging: a new immune-metabolic viewpoint for age-related diseases. Nat Rev Endocrinol. 2018 Oct;14(10):576-590. doi: 10.1038/s41574-018-0059-4. PMID 30046148
- [Background] Krogh J, Benros ME, Jorgensen MB, Vesterager L, Elfving B, Nordentoft M. The association between depressive symptoms, cognitive function, and inflammation in major depression. Brain Behav Immun. 2014 Jan;35:70-6. doi: 10.1016/j.bbi.2013.08.014. Epub 2013 Sep 7. PMID 24016864
- [Background] Borges SM, Radanovic M, Forlenza OV. Correlation between functional mobility and cognitive performance in older adults with cognitive impairment. Neuropsychol Dev Cogn B Aging Neuropsychol Cogn. 2018 Jan;25(1):23-32. doi: 10.1080/13825585.2016.1258035. Epub 2016 Dec 9. PMID 27934540
- [Background] Tang HY, Riegel B, McCurry SM, Vitiello MV. Open-Loop Audio-Visual Stimulation (AVS): A Useful Tool for Management of Insomnia? Appl Psychophysiol Biofeedback. 2016 Mar;41(1):39-46. doi: 10.1007/s10484-015-9308-7. PMID 26294268
- [Background] Tang HY, Vitiello MV, Perlis M, Mao JJ, Riegel B. A pilot study of audio-visual stimulation as a self-care treatment for insomnia in adults with insomnia and chronic pain. Appl Psychophysiol Biofeedback. 2014 Dec;39(3-4):219-25. doi: 10.1007/s10484-014-9263-8. PMID 25257144
- [Background] Derner M, Chaieb L, Surges R, Staresina BP, Fell J. Modulation of Item and Source Memory by Auditory Beat Stimulation: A Pilot Study With Intracranial EEG. Front Hum Neurosci. 2018 Dec 11;12:500. doi: 10.3389/fnhum.2018.00500. eCollection 2018. PMID 30618681
- [Background] Chaieb L, Wilpert EC, Hoppe C, Axmacher N, Fell J. The Impact of Monaural Beat Stimulation on Anxiety and Cognition. Front Hum Neurosci. 2017 May 15;11:251. doi: 10.3389/fnhum.2017.00251. eCollection 2017. PMID 28555100